CLINICAL TRIAL: NCT06103773
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Oral Doses and to Evaluate the Food Effect of TollB-001
Brief Title: A Study of Single and Multiple Oral Doses of TollB-001
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toll Biotech Co. Ltd. (Beijing) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TLBT-TOLLB-001-I
Record Dates: First submitted 2023-09-22; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- SAD-TollB-001 50mg Dosage groups (Experimental): drug：TollB-001 tablets（50mg，single-dose, on the first day）
  Interventions: Drug: TollB-001 tablets; Drug: TollB-001 placebo
- SAD-TollB-001 100mg Dosage groups (Experimental): drug：TollB-001 tablets （100mg，single-dose, on the first day）
  Interventions: Drug: TollB-001 tablets; Drug: TollB-001 placebo
- SAD-TollB-001 200mg Dosage groups (Experimental): drug：TollB-001 tablets （200mg，single-dose, on the first day）
  Interventions: Drug: TollB-001 tablets; Drug: TollB-001 placebo
- SAD-TollB-001 400mg Dosage groups (Experimental): drug：TollB-001 tablets （400mg，single-dose, on the first day）
  Interventions: Drug: TollB-001 tablets; Drug: TollB-001 placebo
- SAD-TollB-001 800mg Dosage groups (Experimental): drug：TollB-001 tablets （800mg，single-dose, on the first day）
  Interventions: Drug: TollB-001 tablets; Drug: TollB-001 placebo
- SAD-TollB-001 1000mg Dosage groups (Experimental): drug：TollB-001 tablets （1000mg，single-dose, on the first day）
  Interventions: Drug: TollB-001 tablets; Drug: TollB-001 placebo
- MAD- TollB-001 100mg Dosage groups (Experimental): drug：TollB-001 tablets （100mg，Multiple-dose, once per day for 5 days）
  Interventions: Drug: TollB-001 tablets; Drug: TollB-001 placebo
- MAD- TollB-001 200mg Dosage groups (Experimental): drug：TollB-001 tablets （200mg，Multiple-dose, once per day for 5 days）
  Interventions: Drug: TollB-001 tablets; Drug: TollB-001 placebo
- MAD-TollB-001 400mg Dosage groups (Experimental): drug：TollB-001 tablets （400mg，Multiple-dose, once per day for 5 days）
  Interventions: Drug: TollB-001 tablets; Drug: TollB-001 placebo
- MAD-TollB-001 800mg Dosage groups (Experimental): drug：TollB-001 tablets （800mg，Multiple-dose, once per day for 5 days）
  Interventions: Drug: TollB-001 tablets; Drug: TollB-001 placebo
- FE-Low Dosage groups (Experimental): drug：TollB-001 tablets（Subjects in the fasting-fed sequence group will be administered with TollB-001 under fasting condition in the first period and under fed condition in the second period; subject in the fed-fasting sequence group will be administered with TollB-001 under fed condition in the first period and under fasting condition in the second period. The two periods of cross-administration will have a washout period of 5-10 days）
  Interventions: Drug: TollB-001 tablets
- FE-High Dosage groups (Experimental): drug：TollB-001 tablets Subjects in the fasting-fed sequence group will be administered with TollB-001 under fasting condition in the first period and under fed condition in the second period; subject in the fed-fasting sequence group will be administered with TollB-001 under fed condition in thefirst period and under fasting condition in the second period. The two periods of cross-administration will have a washout period of 5-10 days）
  Interventions: Drug: TollB-001 tablets

INTERVENTIONS:
Drug: TollB-001 tablets — TollB-001 treatment
  Other Names: TollB-001
Drug: TollB-001 placebo — TollB-001 Placebo
  Arms: MAD- TollB-001 100mg Dosage groups; MAD- TollB-001 200mg Dosage groups; MAD-TollB-001 400mg Dosage groups; MAD-TollB-001 800mg Dosage groups; SAD-TollB-001 1000mg Dosage groups; SAD-TollB-001 100mg Dosage groups; SAD-TollB-001 200mg Dosage groups; SAD-TollB-001 400mg Dosage groups; SAD-TollB-001 50mg Dosage groups; SAD-TollB-001 800mg Dosage groups

SUMMARY:
The primary objective is to evaluate the safety and tolerability of TollB-001 following the administration of single or multiple oral doses in healthy adult subjects

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, PK, and PD of single or multiple dose(s) of TollB-001 administered orally in healthy adult subjects and the food effect on the PK of a single dose of TollB-001 with a randomized, open-label and two-period crossover design.

This study includes three parts. Part A: single ascending dose (SAD) study; Part B: multiple ascending dose (MAD) study; and Part C: FE study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects between the age of 18 and 45 (both inclusive) when signing the informed consent form (ICF)
2. Able to give a signed written ICF (the consent form must be signed by the subject prior to any study-specific procedures); have a full understanding of the study content, procedures, and possible AEs; and be willing and able to comply with study procedures and follow-up examinations
3. Body mass index (BMI, weight [kg]/height2 [m2]) within 19.0-26.0 kg/m2 (both inclusive), with total body weight > 50 kg for male subjects and > 45 kg for female subjects.
4. The subjects must be willing to use efficient physical contraception methods with a contraceptive failure rate of<1% with their reproductive age partners within 90 days from signing the ICF to the last administration of the investigational drug (such as condoms , intrauterine devices)
5. Male subjects must also be willing to refrain from donating sperm for 90 days from the first administration of the investigational drug to the last administration of the investigational drug
6. Results of vital signs, physical examination, laboratory examinations, abdominal and urinary B-ultrasound, 12-lead ECG, and other examination are normal or abnormal but not clinically significant. QT interval corrected for heart rate according to Fridericia's formula (QTcF) must be within the following ranges: QTcF ≤ 450 msec for male subjects, and QTcF ≤ 470 msec for female subjects. Assessment may be repeated if deemed appropriate by the investigator.
7. Ability to swallow all IMPs.

Exclusion Criteria:

Subjects were excluded if they meet any of the following exclusion criteria:

1. Known or suspected allergy or hypersensitivity to any component of TollB-001, known allergic constitution or allergy to two or more foods or drugs.
2. Severe gastrointestinal diseases, such as patients who have undergone major gastrointestinal surgery that would potentially alter absorption and/or excretion of orally administered drugs (except for cholecystectomy, appendectomy, hernia repair), or medical history of ulcer, gastrointestinal bleeding, gastritis, etc.
3. History or clinical manifestations of any clinically significant gastrointestinal, gallbladder or biliary tract, renal, urologic, pulmonary, neurological, cardiovascular, endocrinological, hematological, immunologic, dermatologic, metabolic disorder, or psychiatric disease (as determined by the investigator).
4. Current or chronic history of liver disease or known hepatic ,or clinically significant of biliary abnormalities , or clinically significant abnormal results of liver function test at screening, including alanine amino transferase (ALT) or/and aspartate aminotransferase (AST) > 1.5 × upper limit of normal (ULN)or/and total bilirubin > ULN.
5. eGFR < 90 mL/min/1.73 m2 calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at screening or on Day-1.
6. Current or history of clinically significant cardiac arrhythmias (symptomatic or asymptomatic).
7. Serious infection within 3 months prior to dosing or symptoms of infection within 7 days before dosing, including acute and chronic infections and local infections (bacterial, viral, parasitic, fungal, or other opportunistic pathogens), which is inappropriate to participant as deemed by the investigator.
8. Major illness or surgery within 3 months before dosing ,or planned surgery during the study period.
9. Intolerance to venipuncture.
10. Participation in any clinical study or received any other investigational product or device within 4 weeks prior to the first dose or 5 times the half-life of the specific drug/biologics(whichever is longer), or plan to take an investigational agent during the study.
11. Donated blood > 400 mL or significant blood loss (equivalent to 400 mL), or received blood transfusion within 3 months of prior to screening, or have plans to donate blood during the study.
12. History of malignancy within 5 years prior to screening (excluding non-melanoma skin cancer that has been resected).
13. Positive results of any of the following tests at screening: serum hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV RNA or HCV antibodies [Ab]), human immunodeficiency virus 1 and 2 (HIV)Ab, or Treponema pallidum (TP) Ab.
14. Active tuberculosis (TB) infection indicated by chest radiography orγ-interferon at screening or within 3 months prior to screening. TB test positive, or active or latent TB infection as discretion of the investigator according to clinical practice, or history of TB, or currently receiving treatment for this disease.
15. Plans to receive administration of any live vaccine within 4 weeks before dosing or up to 30 days after the last dose of IMP.
16. Use of drugs, including prescription, over-the-counter medications herbal products, vitamins, and minerals, within 2 weeks prior to the first dose or within 5 times the elimination half-life of the medication prior to first dosing（whichever is longer）.
17. Participated in strenuous exercise from 48 hours prior to Day-1 .
18. Unwilling to refrain from any food or beverage containing caffeine or producing xanthine after metabolism (e.g., tea, coffee, chocolate, cola, red cattle) from 24 hours prior to Day -1 and during the study.
19. Use of food or beverages likely to influence liver metabolism, within 14 days prior to the first dose of the IMP (e.g., star fruit, pomelos, grapefruit, and Seville oranges). Use of any drugs or nutrients known to modulate cytochrome P450 (CYP) 1A2, 2B6, 2C8, 2C9, 2C19, 2D6, 3A and transporter OATP1B1,1B3, OAT3, OCT2 activity (refer to Appendix 3) or any strong or moderate inhibitors or inducers ofCYP1A2, BCRP, OATP1B1, OATP1B3, and OAT3 (refer to Appendix 4) starting from 14 days priorto dose administration on Day 1.
20. History of significant alcohol abuse within 6 months prior to screening or use of more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of alcohol 40% or 150 mL of wine) within 90 days prior to screening or alcohol breath test >0.0mg/100ml at screening, or unwilling to refrain from consumption of alcohol during the study.
21. Use of tobacco or nicotine products or smoking within 90 days (more than 5 cigarettes per day) prior to screening and unwilling to refrain from 24 hours prior to Day -1 and during the study.
22. Drug abuse or those who have taken drugs (such as cocaine, phencyclidine, etc.) within one year prior to screening (consultation); Or those who are positive for urine drug abuse screening (methamphetamine, ketamine, MDMA ,tetrahydrocannabinoid acid, morphine) during screening.
23. Women who are lactating or positive pregnancy test within at screening or during the study period, or planning to become pregnant during the study period.
24. Acute illness occurs or concomitant medication required from screening to dosing.
25. Constipated or irregular bowel movements.
26. Any other situation that researchers believe may affect the subject's ability to provide informed consent or follow the trial protocol, or the subject's participation in the trial may affect the trial results or their own safety.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-06-09 (Estimated); Study Completion 2024-06-09 (Estimated)

PRIMARY OUTCOMES:
Red blood cell count(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  Red blood cell count
hematocrit(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  hematocrit
hemoglobin(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  hemoglobin
white blood cell count(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  white blood cell count
whiteblood cell differential count(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  whiteblood cell differential count
plateletcount(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  plateletcount
Alanine aminotransferase(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  Alanine aminotransferase
aspartateaminotransferase(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  aspartateaminotransferase
alkaline phosphatase(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  alkaline phosphatase
gamma-glutamyl transpeptidase(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  gamma-glutamyl transpeptidase
total bilirubin(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  total bilirubin
direct bilirubin(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  direct bilirubin
blood ureanitrogen (or blood urea)(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  blood ureanitrogen (or blood urea)
creatinine(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  creatinine
glucose(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  glucose
total protein(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  total protein
creatine kinase(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  creatine kinase
Activated partial thromboplastin time(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  Activated partial thromboplastin time
prothrombin time(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  prothrombin time
internationalnormalized ratio(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  internationalnormalized ratio
fibrinogen(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  fibrinogen
urine pH(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  urine pH
urine specific gravity(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  urine specific gravity
urine glucose(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  urine glucose
urine protein(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  urine protein
urobilinogen(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  urobilinogen
urine bilirubin(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  urine bilirubin
urine leukocyte(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  urine leukocyte
urine ketone body(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  urine ketone body
urine red blood cells(physiological parameter) by investigator | Baseline（Screening）up to last follow-up visit(SAD:Screening up to Week 1;MAD:Screening up to Week 2;FE:Screening up to Week 2 plus 10 days)
  urine red blood cells
AE/SAE monitoring by ToxicityGrading Scale for Healthy Adults and Volunteers Enrolled in Preventative Vaccine Trials,2007 (70 FR 22664) | First dose up to last follow-up visit（for a maximum of 20 days）
  AE/SAE monitoring
physical examination(physiological parameter) by investigator | First dose up to last follow-up visit（for a maximum of 20 days）;SAD:Screening,Day2,Day5 or ET Visit;MAD:Screening,Day3,Day6,Day9 or ET Visit;FE:Screening,Period 1 Day2,Period 1 Day5;Period 2 Day-1,Period 2 Day2,Period 2 Day5 or ET Visit.
  The assessments of general appearance, head(including ears, eyes, nose, throat), neck, skin, cardiovascular system, respiratory system,abdominal system, nervous system, musculoskeletal system, and lymphatic system
blood pressure(systolic pressure and diastolic pressure)(physiological parameter) by investigator | For a maximum of 20 days;SAD:Screening,Day1 to Day5 or ET Visit;MAD:Screening,Day1 to Day9 or ET Visit;FE:Screening,Period 1 Day1 to Day5;Period 2 Day-1 to Day5 or ET Visit.
  blood pressure(systolic pressure and diastolic pressure)
pulse(physiological parameter) by investigator | For a maximum of 20 days;SAD:Screening,Day1 to Day5 or ET Visit;MAD:Screening,Day1 toDay9 or ET Visit;FE:Screening,Period 1 Day1 to Day5;Period 2 Day-1 to Day5 or ET Visit.
  pulse
respiratory rate(physiological parameter) by investigator | For a maximum of 20 days;SAD:Screening,Day1 to Day5 or ET Visit;MAD:Screening,Day1 toDay9 or ET Visit;FE:Screening,Period 1 Day1 to Day5;Period 2 Day-1 to Day5 or ET Visit.
  respiratory rate
body temperature(physiological parameter) by investigator | For a maximum of 20 days;SAD:Screening,Day1 to Day5 or ET Visit;MAD:Screening,Day1 toDay9 or ET Visit;FE:Screening,Period 1 Day1 to Day5;Period 2 Day-1 to Day5 or ET Visit.
  body temperature
12-lead ECGs | For a maximum of 20 days;SAD:Screening,Day1 to Day5 or ET Visit;MAD:Screening,Day1 to Day9 or ET Visit;FE:Screening,Period 1 Day1,Period 1 Day3,Period 1 Day5;Period 2 Day-1,Period 2 Day1,Period 2 Day3,Period 2 Day5 or ET Visit.
  ECGs done in triplicate; heart rate, PR interval, QT and QTc interval and QRS duration
B-ultrasound(physiological parameter) by investigator | For a maximum of 20 days;SAD:Screening,Day5 or ET Visit;MAD:Screening,Day9 or ET Visit;FE:Screening,Period 1 Day5;Period 2 Day5 or ET Visit.
  liver, gallbladder, spleen, pancreas, kidney and bladder

CONTACTS AND LOCATIONS:
Overall Officials: wen he, Study Director — Chengdu Fifth People's Hospital
Locations (1):
- Chengdu Fifth People's Hospital, Chengdu, Sichuan, China